CLINICAL TRIAL: NCT07013357
Title: Digital, Community-Advised, Social Action Cluster-Randomized Trial to Increase Civic Participation and Social Connection in the US
Brief Title: Community Discussions and Social Participation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 856943
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Social Connectedness; Community Engagement; Physical Wellbeing
Keywords: Virtual Intervention; Setting Goals; Civic Participation; Social Connection; Physical Well-being; Anxiety and Distress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Cohorts will be randomized to the experimental or control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention sessions along with GROV engagement (Experimental): Participants in the experimental group will attend three highly structured Virtual intervention sessions, hosted on Zoom and facilitated by trained research team members. They will also be encouraged to sign up for GROV after completing the baseline and are expected to engage with the GROV platform throughout the study period. The GROV platform will serve as a digital community space for ongoing interaction and discussion.
  Interventions: Behavioral: Virtual Community Intervention
- Self-help sessions without GROV engagement (Active Comparator): Participants will attend loosely structured, self-run, virtual group self-help sessions at the same time and duration as intervention sessions. No discussion on the GROV platform for the control group.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Virtual Community Intervention — Participants will attend three Virtual intervention sessions, hosted on Zoom and facilitated by trained research team members. Co-facilitators (comprised of lab staff) will also be there to ensure no technical difficulties and record the meeting. Sessions will be held at the same time each week for three weeks. After each session, facilitators will be assessed for fidelity based on feedback from the session quality assessment survey.
  Every session will have its primary focus, respectively:
  Session 1 will focus on fostering social connections. Session 2 will focus on setting mental/physical wellbeing goals. Session 3 will focus on pursuing similar goals for their community.
  During the sessions, participants will work together and offer mutual support under the direction of the facilitator. Furthermore, facilitators will communicate with participants between sessions to check in on their progress toward their goals.
  Arms: Intervention sessions along with GROV engagement
Behavioral: Control — Participants will attend three 90-minute Virtual self-help sessions, hosted on Zoom. Sessions will be held at the same time each week for three weeks, in parallel to the experimental condition. First, the co-facilitator will let participants into the Zoom room and begin the recording. After they introduce themselves, they will remain on mute/camera off for the entire meeting to handle technical difficulties or intervene when violations occur, for example, using inappropriate language. Co-facilitators may also interact with participants through the chat to provide referrals. Then, the discussion leader will explain their role and ask everyone to introduce themselves. As a group, they will set some ground rules. Then, the discussion leaders will guide the discussion, using the Self-Help Session Manual as a reference, which provides structure and reference questions to facilitate discussion. Beyond this guideline, participants can discuss anything they decide as a group.
  Arms: Self-help sessions without GROV engagement

SUMMARY:
This study evaluates a virtual program designed to boost the physical well-being goals, civic engagement, social connection, and anxiety of U.S. adults.

DETAILED DESCRIPTION:
This single-blind, cluster randomized controlled trial aims to develop a virtual intervention designed to support US adults who wish to work with others to achieve physical wellbeing goals, improve social connectedness, promote community engagement, and reduce anxiety. Research coordinators randomize 10 participants to facilitator-led intervention sessions, and 10 to self-run discussion sessions by assigning random computer generated codes, sorting in ascending order, and alternating "control" and "experimental" assignments. This project is funded by the Annenberg Endowment of the Division of Communication Science.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Residency: Must live in a U.S. state (including D.C. and U.S. territories)
* Technology access: Reliable internet, a webcam, and Zoom capability in a private space
* Language: Able to read and speak English (all materials and sessions are in English)

Exclusion Criteria:

* Inability to provide informed consent
* Under 18 years of age
* Not living in the U.S.
* Lack of reliable access to the required technology (e.g., internet-connected device)
* Unable to read and understand English at the level required for full participation in the study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Physical Wellbeing Goal Progress | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  How much progress have you made towards this goal? (1, No progress | 2, Little progress | 3, Some progress | 4, Substantial progress | 5, Goal achieved)
Civic Participation | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  In the past month (baseline)/since the beginning of this study (follow-up) have you participated in or taken action through a group or organization to improve yourself, your community, or help others? (0, No | 1, Yes)
Social Connection | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  In the past month (baseline)/Since joining the study (follow-up), have you started a new social connection or re-established an old one? (0, No | 1, Yes)
Anxiety | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  On a scale from 1, None of the time | 2, A little of the time | 3, Some of the time | 4, Most of the time | 5, All of the time ...
  * In the past month (Baseline)/Since joining the study, about how often did you feel anxious?
  * In the past month (Baseline)/Since joining the study, about how often did you feel restless or fidgety?
  * In the past month (Baseline)/Since joining the study, about how often did you feel that everything took effort?
  * In the past month (Baseline)/Since joining the study, about how often did you feel so sad that nothing could cheer you up?
  Mean of 4 item raw score.

SECONDARY OUTCOMES:
Attitude toward Health | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  I feel confident in my ability to seek help for my health problems. I feel confident in my ability to solve my health problems. I feel comfortable with challenges related to solving my health problems.
  Response Scale: 1, Not confident at all | 2, Slightly | 3, Somewhat | 4, Confident | 5, Very confident Score: Mean of 1-5 Scores
Attitude toward Social Connections | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  How easy is it to get help from members of your community if you need it? 1, Impossible | 2, Difficult | 3, Possible | 4, Easy | 5, Very easy How often do you feel that there are people you can turn to? 1, Never | 2, Sometimes | 3, Often | 4, Most of the time | 5, Always To what extent were you hesitant to tell others what you want or need from them? 1, Very much | 2, Quite a bit | 3, Somewhat | 4, A little | 5, Not at all To what extent are you willing to seek support from others if you need it? 1, Not at all | 2, A little | 3, Somewhat | 4, Quite a bit | 5, Very much When you feel afraid, anxious, or uncertain, how often do you seek help or support from others in your life (e.g., reaching out to neighbors, joining support groups, attending social events?) 1, Never | 2, Sometimes | 3, Often | 4, Most of the time | 5, Always
  Score: Mean of 1-5 Scores
Political Trust | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  How much can you trust the federal government to do what is right regarding the social changes you want to make? (1, No trust | 2, Little | 3, Some | 4, Quite a lot | 5, A great deal ) How often can you trust your state government to do what is right when it comes to handling the social changes you want to make? (1, Never | 2, Rarely | 3, Sometimes | 4, Often | 5, Always ) How often can you trust your local government to do what is right when it comes to handling the social changes you want to make? (1, Never | 2, Rarely | 3, Sometimes | 4, Often | 5, Always )
  Score: Mean of 1-5 scores
Attitude toward Political Participation | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  How likely or unlikely are you to vote in the next local, state, or national elections? (1, Extremely unlikely | 2, Unlikely | 3, Neutral | 4, Likely | 5, Extremely likely)
Attitude toward Problem Solving | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  When I face problems, I am confident that I can solve them. How confident do you feel in your ability to achieve your goals? How comfortable are you with taking on new challenges? Response Scale: 1, Almost never | 2, Rarely | 3, Sometimes | 4, Often | 5, Almost always Score: Mean of 1-5 Scores
Attitude toward Civic Engagement | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  I feel responsible for the well-being of others in groups I belong to I am committed to help others in groups I belong to I believe that all citizens have a responsibility to their fellow citizens I believe that it is important to be informed of societal issues Response Scale: 1, Strongly disagree | 2, Disagree | 3, Neither | 4, Agree | 5, Strongly agree In the past month (Baseline)/Since the beginning of the study (follow-up), how concerned, if at all, were you about others with whom you are connected? Response Scale: 1, Not at all | 2, Slightly | 3, Moderately | 4, Very | 5, Extremely Score: Mean of 1-5 Scores

OTHER OUTCOMES:
Exploratory Outcome: Wellbeing | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  On a scale from1, None of the time | 2, A little of the time | 3, Some of the time | 4, Most of the time | 5, All of the time
  * In the past month (baseline)/Since joining the study (follow-up), I have felt cheerful and in good spirits.
  * In the past month (baseline)/Since joining the study (follow-up), I have felt calm and relaxed.
  * In the past month (baseline)/Since joining the study (follow-up), I have felt active and vigorous.
  * In the past month (baseline)/Since joining the study (follow-up), I woke up feeling fresh and rested.
  * In the past month (baseline)/Since joining the study (follow-up), my daily life has been filled with things that interest me.
  Score: Mean of 5 item raw scores
Exploratory Outcome: Social Support | Measured at Baseline and Immediate Follow-Up (1 week after the last session)
  On a scale from 1, None of the time | 2, A little of the time | 3, Some of the time | 4, Most of the time | 5, All of the time ...
  * Since joining the study, how often do you feel that you are "in tune" with the people around you?
  * (rev) Since joining the study how often do you feel that you lack companionship?
  * (rev) Since joining the study, how often do you feel isolated from others?
  * Since joining the study, how often do you feel that there are people you can turn to?
  Score: Mean of 4 item raw scores. (rev) means reverse scored.

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Albarracin, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT07013357/Prot_SAP_001.pdf